CLINICAL TRIAL: NCT05880680
Title: SEAL™ME: Saccular Endovascular Aneurysm Lattice System Multicenter Enrollment Global Registry
Acronym: SEAL™ME
Status: Recruiting | Type: Observational
Sponsor: Galaxy Therapeutics INC (Industry)
Responsible Party: Sponsor
Other Study IDs: TP0050
Record Dates: First submitted 2023-05-19; First posted 2023-05-30 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Aneurysm; Aneurysm, Ruptured
MeSH Terms: conditions — Aneurysm; Aneurysm, Ruptured

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: SEAL Device — Using standard interventional endovascular techniques, the device is navigated via the push wire delivery system through compatible neurovascular microcatheters to the aneurysm lumen or target site. The device is positioned into its target aneurysm lumen and is electrically detached by the operator with a hand-held, battery-powered detachment handle designed specifically for the SEAL Embolization System.

SUMMARY:
Prospective, international, single-arm, multicenter, registry study. Patients presenting with evidence of Wide Neck unruptured or ruptured intracranial aneurysm (≤ 20 mm in widest diameter) requiring treatment will be enrolled into the study and treated using the SEAL™ System.

DETAILED DESCRIPTION:
Prospective, international, single-arm, multicenter, registry study. Patients presenting with evidence of Wide Neck unruptured or ruptured intracranial aneurysm (≤ 20 mm in widest diameter) requiring treatment will be enrolled into the study and treated using the SEAL™ System. Immediate post-procedure angiographic findings, clinical presentation, safety, and optional imaging follow-up for each subject will be collected at 24 hours or discharge, 3 months, 6 months, and required primary end point 12 months post-procedure. DSA at 12 months will be required imaging for the primary effectiveness endpoint assessment. Subjects follow up will continue annually for a total of five years post procedure.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 80 years of age at the time of screening.
2. Unruptured aneurysm requiring endovascular treatment suitable for SEAL device and meet the AHA guidelines for management of unruptured aneurysm.5 If there is evidence of an additional aneurysm requiring treatment, the secondary aneurysm must also be treatable using a SEAL™ System Device, either during a single procedure or consecutive procedures.

   No additional preplanned implanted devices are permissible except for as medically required for patient safety during the procedure.
3. Ruptured aneurysm

   1. Ruptured aneurysms may be included according to the following criteria: The subject is neurologically stable with no seizure at the onset of the SAH, not requiring EVD placement prior to inclusion.
   2. Hunt and Hess scale of 3 or less at the time of treatment.
   3. Modified Disability Scale (mRS) of ≤2 prior to presentation or aneurysm rupture.
   4. Meet the AHA guidelines for management of ruptured aneurysm.6
4. The index intracranial aneurysm (IA) to be treated must include the following features:

   1. Aneurysm features suitable for endovascular treatment with an intrasaccular device per the treating interventionist.
   2. Saccular morphology.
   3. Located at a bifurcation, terminus, or sidewall in the anterior or posterior circulation.
   4. 2.5 mm-20 mm in dome diameter.
   5. Wide-neck aneurysm with neck size ≥ 4mm or Dome-to-Neck (DN) ratio < 2.
5. Aneurysm treatment does not require the preplanned use of any additional implanted devices.
6. Subject is able to maintain compliance with all aspects of screening, evaluation, treatment, and post-procedure follow-up schedule.
7. Baseline pre-procedure mRS of 0-2 for unruptured aneurysm and 0-2 prior to the SAH for the ruptured aneurysms.
8. Ability to obtain written informed consent from subject or legally authorized representative in SAH subjects prior to the initiation of any study procedures.

Exclusion Criteria:

1. Aneurysm features unsuitable for endovascular treatment with an intrasaccular device such as fusiform, dissecting pseudo aneurysm, or mycotic aneurysm.
2. Aneurysms smaller than 2.5 mm and larger than 20 mm in dome width.
3. Inability to access target aneurysm with microcatheter due to intracranial atherosclerosis, proximal or intracranial vessel tortuosity or poor aneurysm angle take-off.
4. Patients with two 360 degrees loops in the carotid or vertebral arteries.
5. Presence of vascular disease or other vascular abnormality that could prohibit access to index aneurysm such carotid stenosis or diminished caliber of the target artery.
6. Clinical, angiographic, or CT evidence of CNS arterial vasculitis, Moyamoya disease, intracranial tumor (except small meningioma), or any other intracranial vascular malformations.
7. Patients with high risk for recurrent ischemic stroke due to previous history of ischemic stroke symptoms such as transient ischemic attacks (TIAs), minor, or major strokes within the past 60 days. Other stroke risk factors such as intracranial stenosis or atrial fibrillation.
8. Patients with hemodynamic or medical compromise due to medical comorbidities such as severe unstable congestive heart failure (ejection fraction <30%) or severe COPD requiring home oxygen.
9. Modified Rankin Scale (mRS) score of > 2 prior to presentation.
10. Target index aneurysm that has been previously treated and contains devices, implants, or coils that could interfere with correct SEAL™ device placement.
11. Subject is pregnant or a lactating female (For females of child-bearing potential, a positive pregnancy test within 7 days of the day of procedure or refusal to use a medically accepted method of birth control for the duration of the study.
12. Currently on anticoagulation therapy or has a known blood dyscrasia, coagulopathy, or hemoglobinopathy.
13. Currently enrolled in another investigational study or post-market study that could affect the safety and efficacy of aneurysm treatment or interfere with the study follow-up schedule.
14. Presence of an acute life-threatening illness requiring treatment.
15. Life expectancy of <1 year.
16. Subject has an uncontrolled co-morbid medical condition, that would adversely affect participation in the study.
17. Patient with chronic kidney disease (and not on dialysis) with creatinine > 2.0.
18. Subject is a prisoner or member of other vulnerable population.
19. Subject that is in the opinion of the treating interventionalist is not suitable for the study.

    * Sensitivity to nickel is not specifically excluded, Galaxy Therapeutics, Inc (GTI) performed ASTM F2129 testing recommended by the FDA in its 2015 and 2019 guiding documents. GTI results from the testing indicated that SEALTM meets the acceptance criteria that there is a high probability that the margin of safety against pitting (Eb-Er) is 200mV or higher, therefore, with high confidence, no further testing is required. The IFU contains the following precaution: "For patients with known hypersensitivity or allergic reaction to the implant components such as titanium or to nickel, use of the SEALTM System may lead to allergic reaction and user should counsel the patient on the device components".

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult subjects between 20 and 80 years of age and presenting with an unruptured or ruptured saccular Wide Neck intracranial aneurysm with less or equal to 20 mm in its widest diameter (2.5mm-20mm range) that in the opinion of the Principal Investigator requires treatment and suitable candidate for intrasaccular flow diversion treatment, who meet all eligibility criteria, will be considered for study enrollment. Up to 200 adult subjects will be enrolled in the study in up to 25 centers.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2030-06-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with successful aneurysm occlusion at 12 months without parent artery stenosis or retreatment, as determined by independent core lab. | 12 Months
  * Index aneurysm occlusion is defined as achieving WEB Occlusion Scale (WOS) of A or B at 12 months.1,2
  * Index aneurysm parent arterial stenosis is defined as diameter stenosis of >50%.
  Index aneurysm retreatment at any point post procedure throughout the duration of the study period will be considered a failure for the primary efficacy endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Osama Zaidat, MD, MS, Study Chair — Mercy Health, OH
Locations (4):
- Angiosur, Itagüi, Medellín, Colombia
- Auckland City Hospital, Auckland, Auckland, New Zealand
- Punjab Institute of Neuroscience (PINS), Lahore, Lahore, Pakistan
- Hospital Universitari Vall d'Hebron, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No